CLINICAL TRIAL: NCT01322607
Title: Task-oriented Training for Stroke: Impact on Function Mobility
Acronym: TOTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: O7194-W
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Cerebrovascular Accident; Stroke
Keywords: Exercise; Rehabilitation; Stroke
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: High-Intensity Program (Other): High-intensity treadmill-based exercise
  Interventions: Behavioral: High-intensity Treadmill Exercise
- Arm 2: Low-Intensity Program (Other): Low-intensity lifestyle intervention (group exercise)
  Interventions: Behavioral: Low-intensity Lifestyle Intervention

INTERVENTIONS:
Behavioral: High-intensity Treadmill Exercise — High-intensity treadmill walking program
  Arms: Arm 1: High-Intensity Program
Behavioral: Low-intensity Lifestyle Intervention — A low-intensity lifestyle intervention targeted towards group exercises incorporating balance, coordination, and strength.
  Arms: Arm 2: Low-Intensity Program

SUMMARY:
Residual neurological deficits from stroke lead to gait inefficiencies, resulting in an extremely high energy cost of movement and contributing to overall disability and lower quality of life. Therefore, interventions targeting movement economy should be developed for those in the chronic phase of stroke recovery. This study is designed to compare the effect of two distinctly different exercise paradigms (a higher-intensity treadmill training program and a lower-intensity group exercise program) on economy of movement during over-ground walking and activities of daily living, as well as the extent to which gains in muscular strength, muscular endurance, and balance predict changes in movement economy.

ELIGIBILITY:
Inclusion Criteria:

* Stroke > 6 months prior with residual hemiparetic gait in women or men aged 40-85 years.
* Completion of all regular post-stroke physical therapy
* Adequate language and neurocognitive function to participate in testing and training and to give adequate informed consent.
* Able to rise from a chair unaided.
* Able to walk 10 meters without human assistance.

Exclusion Criteria:

* Regular structured aerobic exercise (> 2x week).
* Alcohol consumption > 3 oz. liquor, or 3 x 4 oz glasses of wine, or 3 x 12 oz. beers per day, by self-report.
* Clinical history of

  * unstable angina,
  * recent (< 3 months) myocardial infarction or congestive heart failure (NYHA category II),
  * hemodynamically significant valvular dysfunction,
  * Peripheral Arterial Obstructive Disease with claudication,
  * major orthopedic, chronic pain, or non-stroke neuromuscular disorders restricting exercise,
  * pulmonary or renal failure,
  * poorly controlled hypertension (>190/110), measured on at least two separate occasions
  * recent hospitalization for severe disease or surgery
  * severe or global receptive aphasia which confounds reliable testing and training.
* Untreated major depression as documented by a Center for Epidemiological Studies-Depression score of >16 and confirmed by clinical interview.
* Pregnancy.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa D Stookey, PhD MS, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Liu X, Zhang Y, Li F, Liu L, Du J, Song WQ. Test-retest reliability and practice effects of shape trail test in stroke patients. Top Stroke Rehabil. 2025 Oct;32(7):779-788. doi: 10.1080/10749357.2025.2457282. Epub 2025 Mar 13. PMID 40079581
- [Derived] Stookey AD, Macko RF, Ivey FM, Katzel LI. Evaluating Test-Retest Reliability of Fatigability in Chronic Stroke. J Stroke Cerebrovasc Dis. 2021 Sep;30(9):105895. doi: 10.1016/j.jstrokecerebrovasdis.2021.105895. Epub 2021 Jul 7. PMID 34242857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hemiparetic stroke survivors (>6 months) with residual hemiparetic gait in women/men aged 30-85 years who completed all therapy were recruited. They had to have adequate language and neurocognitive function, give adequate informed consent, able to rise from a chair unaided, and able to walk 10 meters without human assistance.
Period: Overall Study
Arm/Group | Arm 1: High-Intensity Program | Arm 2: Low-Intensity Program
Started | 11 | 9
Completed | 10 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: High-Intensity Program | Arm 2: Low-Intensity Program | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.36 (8.63) | 61.89 (9.03) | 60.5 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 6 | 15
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.57 (5.73) | 30.34 (7.53) | 29.92 (6.43)
Weight [Mean (Standard Deviation); unit: kg] | 88.92 (22.27) | 86.56 (19.57) | 87.86 (20.59)
Height [Mean (Standard Deviation); unit: cm] | 172.79 (10.83) | 169.54 (11.87) | 171.33 (11.13)

OUTCOME MEASURES:

1. Primary Outcome: Economy of Gait
Description: Over-ground gait economy measured using a portable metabolic monitoring system, K4b2 during a 6 minute walk, with subjects walking at their comfortable self-selected walking speed while open circuit spirometry collects break-by-break data. The K4b2 consists of a small battery pack and portable gas analyser (weighing less than 1 kg) that participants wear on their chest. Attached to the portable system is a flexible rubber facemask with flowmeter used for breath-by-breath analysis. The mean rate of oxygen consumption (VO2) will be calculated based on the final 3 minutes of a 6-minute walk under steady state oxygen consumption conditions. A 6 minute walk is a distance most representative of community-based ambulatory capacity and is a sensitive outcome measure in exercise studies in chronic stroke subjects. The higher the VO2 used during the 6 minute walk, represents a less efficient economy of gait.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Arm 1: High-Intensity Program | Arm 2: Low-Intensity Program
Number analyzed (Participants) | 10 | 9
ml/kg/min | 13.44 (3.15) | 12.67 (3.51)

2. Secondary Outcome: Muscular Strength
Description: Strength measured by torque of isokinetic maximal concentric knee extensor volitional contractions of paretic and non-paretic leg at multiple angular velocities (30, 90, and 120°/sec). The higher the number the higher the muscular strength. Also performed on resistance equipment for both the Leg Press and Leg Extension. The higher the number the stronger a person is.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: newtons (N)
Arm/Group | Arm 1: High-Intensity Program | Arm 2: Low-Intensity Program
Number analyzed (Participants) | 10 | 9
newtons (N)
  Leg Extension Non-Paretic Leg | 151.82 (53.73) | 113.33 (61.24)
  Leg Extension Paretic Leg | 101.36 (55.64) | 70.0 (35.18)
  Leg Press Non-Paretic Leg | 491.82 (217.42) | 463.33 (146.03)
  Leg Press Paretic Leg | 371.82 (229.78) | 295.56 (170.67)

3. Secondary Outcome: Muscular Endurance
Description: Muscular endurance performed on Leg Press and assessed by a force transducer, while seated. The longer the amount of time participant can maintain a force the better their muscular endurance.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Arm 1: High-Intensity Program | Arm 2: Low-Intensity Program
Number analyzed (Participants) | 10 | 9
seconds
  Leg Press Non-Paretic Leg | 67.55 (24.66) | 67.22 (24.96)
  Leg Press Paretic Leg | 41.63 (22.36) | 40.10 (28.12)

4. Secondary Outcome: Balance
Description: Dynamic Gait Index - another measure related to balance and general function. It includes items of walking while changing speed, turning the head, pivot turning, walking over and around obstacles, and stair climbing. This index ranges from 0 - 24, with 24 representing a high level of balance and general function (the higher the score the better the balance).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: High-Intensity Program | Arm 2: Low-Intensity Program
Number analyzed (Participants) | 11 | 9
units on a scale | 17.01 (4.13) | 14.22 (3.56)

ADVERSE EVENTS:
Time Frame: Adverse event information was obtained for participants for the duration of their time in this study (0-3months)
Arm/Group | Arm 1: High-Intensity Program | Arm 2: Low-Intensity Program
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/9
Other Adverse Events (participants affected / at risk) | 6/11 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: High-Intensity Program (N=11) | Arm 2: Low-Intensity Program (N=9)
Esophagitis/Upper Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant hospitalized for esophagitis/Upper Gastrointestinal Bleed. Proton Pump inhibitor added to medication; eventually cleared by Primary Care Physician to resume participation in the study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: High-Intensity Program (N=11) | Arm 2: Low-Intensity Program (N=9)
Fall (General disorders) | 6 (12) | 8 (14) — All adverse events other than the one serious event reported were participant falls (expected in this population). No serious injuries reported from falls and all falls were due to losing balance (not fainting or loss of consciousness).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes